CLINICAL TRIAL: NCT06447116
Title: An EFS to Evaluate the Safety and Preliminary Effectiveness of the CGuard Prime™ Carotid Stent Placement in the Procedure Setting of Acute Ischemic Stroke.
Brief Title: An EFS to Evaluate the CGuard Prime™ Carotid Stent in Acute Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobs institute (Other)
Responsible Party: Principal Investigator, Adnan Siddiqui, Principal Investigator, Jacobs institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSPIREMD CIP 004
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- C Guard Arm (Experimental)
  Interventions: Device: CGuard Prime™ Carotid Stent System

INTERVENTIONS:
Device: CGuard Prime™ Carotid Stent System — CGuard Prime™ Carotid Stent System

SUMMARY:
The Jacobs Institute is conducting a Sponsor Investigator study of patients ≥ 18 years to establish safety and preliminary effectiveness in treating extracranial stenosis with the CGuard Prime™ Carotid Stent in the setting as an acute ischemic stroke.

DETAILED DESCRIPTION:
A prospective, single-arm, open-label, nonblinded EFS to assess the safety and preliminary effectiveness of the CGuard Prime™ Carotid Stent in adults (18 years of age or older) with extracranial stenosis in the setting as an acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18-year-old; Carotid stenosis with at least ≥ 50% stenosis; National Institute of Health Stroke Scale (NIHSS) >/=6; and evidence of large vessel occlusion (LVO) in the anterior circulation (i.e., intracranial internal carotid artery, M1 and proximal M2) by computed tomography angiography (CTA).

Exclusion Criteria:

* Cannot provide consent or legally authorized representative not available to provide consent. Evidence of intracranial hemorrhage on non-contrast CT or MRI; ASPECTS<6; and any contraindication to dual antiplatelet therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with mRS ≤ 2 at 90 days | 90 days
  Proportion of subjects with mRS ≤ 2 at 90 days

SECONDARY OUTCOMES:
Rate of TICI 2b or greater; Proportion of subjects with sICH within 24 hours; and New stroke within the same territory within 7 days. | 7 days
  Rate of TICI 2b or greater; Proportion of subjects with sICH within 24 hours; and New stroke within the same territory within 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS LOUIS PENA, PhD, Study Director — Jacobs institute
Locations (1):
- Jacobs Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No